CLINICAL TRIAL: NCT02669186
Title: Effects of Anesthetic Technique on Natural Killer Cell Population and Cytotoxicity
Brief Title: Effects of Anesthetic Technique on NK Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Program Director, Anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00039201-1
Record Dates: First submitted 2015-10-06; First posted 2016-02-01 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pain; Anesthesia; Cancer
Keywords: analgesia; cancer; natural killer cell; opioid
MeSH Terms: conditions — Pain; Neoplasms; Agnosia | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Bupivacaine + Fentanyl' (Opioid Group) (Experimental): Group 1 (opioid group) will receive general endotracheal anesthesia augmented with an epidural. The epidural solution intraoperatively and post-operatively will contain fentanyl + bupivacaine titrated to appropriate surgical conditions and post-operative pain control.
  Interventions: Drug: Bupivacaine + Fentanyl
- Bupivacaine (Local Anesthetic Group) (Active Comparator): Group 2 (local anesthetic group) will receive general endotracheal anesthesia augmented with an epidural. The epidural solution intraoperatively and post-operatively will contain bupivacaine titrated to appropriate surgical conditions and post-operative pain control.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine + Fentanyl — General endotracheal anesthesia augmented with an epidural. The epidural solution intraoperatively and post-operatively will contain fentanyl + bupivacaine titrated to appropriate surgical conditions and post-operative pain control.
  Other Names: Sublimaze
  Arms: 'Bupivacaine + Fentanyl' (Opioid Group)
Drug: Bupivacaine — General endotracheal anesthesia augmented with an epidural. The epidural solution intraoperatively and post-operatively will contain bupivacaine titrated to appropriate surgical conditions and post-operative pain control
  Arms: Bupivacaine (Local Anesthetic Group)

SUMMARY:
The proposed study is a pilot prospective, single-blinded, randomized controlled trial evaluating the effects of two routine, standard-of-care, anesthetic techniques on natural killer cell population size and cytotoxicity in patients undergoing exploratory abdominal laparotomies.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years old of either gender
* Diagnosis of abdominal tumor scheduled for exploratory laparotomy with study surgeon
* Must be able to have an epidural

Exclusion Criteria:

* ASA IV and above
* Intolerance, allergy, or contraindication to use of either fentanyl or bupivacaine.
* Significant coronary artery disease (abnormal stress test, myocardial infarction within the last 3 months)
* Uncontrolled hypertension (BP > 140/90)
* Cardiac arrhythmias particularly prolonged QT syndrome
* Drugs known to cause prolonged qT: class IA antiarrhythmics (quinidine, procainamide, dysopyramide), class III antiarrhythmics (sotalol, dofetalide, ibutalide, amiodarone), haloperidol, thioridazine, arsenic trioxide, HIV protease inhibitors, tricyclic antidepressants
* Individuals with significant psychological disorders including: schizophrenia, mania, bipolar disorder or psychosis
* Pregnant or lactating women
* Morbid obesity (BMI > 40 kg/m2) AND/OR weight > 150 kg
* Chronic renal failure ( creatinine > 2.0 mg/dL)
* Liver failure e.g., active cirrhosis
* Alcohol or substance abuse within in the past 3 months
* Uncorrected hypokalemia, hypomagnesemia, hypocalcemia (can be due to diuretics, mineralocorticoid use, laxatives)
* Neuropathic pain
* Chronic opioid consumption (>30mg oxycodone or greater per day)
* Cachexia from any cause
* Systemic use of corticosteroids for greater than 2 weeks in the 6 months prior to surgery
* HIV or other immunosuppressive condition
* Preoperative INR > 1.4 or platelet count < 100
* Sepsis or overlying skin cellulitis at epidural catheter insertion site
* Inability to tolerate/unwillingness to have an epidural catheter for intraoperative/postoperative pain control for any reason, including prior back surgery resulting in distorted anatomy that precludes neuraxial anesthesia.
* Inability to tolerate an epidural solution of either fentanyl or bupivacaine or needs another form of specialized pain control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Natural Killer Cell Cytotoxicty | One Year
  Cytotoxicity will be assessed using Flow Cytometric analysis of cell receptor expression.

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Program Director, Department of Anesthesiology
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buckley A, McQuaid S, Johnson P, Buggy DJ. Effect of anaesthetic technique on the natural killer cell anti-tumour activity of serum from women undergoing breast cancer surgery: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i56-62. doi: 10.1093/bja/aeu200. Epub 2014 Jul 9. PMID 25009196
- [Background] Beilin B, Shavit Y, Hart J, Mordashov B, Cohn S, Notti I, Bessler H. Effects of anesthesia based on large versus small doses of fentanyl on natural killer cell cytotoxicity in the perioperative period. Anesth Analg. 1996 Mar;82(3):492-7. doi: 10.1097/00000539-199603000-00011. PMID 8623949
- [Background] Cata JP, Bauer M, Sokari T, Ramirez MF, Mason D, Plautz G, Kurz A. Effects of surgery, general anesthesia, and perioperative epidural analgesia on the immune function of patients with non-small cell lung cancer. J Clin Anesth. 2013 Jun;25(4):255-62. doi: 10.1016/j.jclinane.2012.12.007. Epub 2013 May 7. PMID 23659826